CLINICAL TRIAL: NCT01000389
Title: A Clinical Trial of the Optimal Treatment Period and Long-term Efficacy of Functional Electrical Stimulation (FES) on Sleep Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medotech A/S (Industry)
Responsible Party: Pernille Wendelboe, Medotech A/S
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMD-02
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Temporomandibular Disorder; Headache
MeSH Terms: conditions — Temporomandibular Joint Disorders; Headache | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Grindcare® (Biofeedback) — Active treatment with functional electrical stimulation

SUMMARY:
To investigate the effect of the treatment with Grindcare® on the parafunction of the muscles- and jaw activity (Bruxism) during sleep.

ELIGIBILITY:
Inclusion Criteria:

* RDC-TMD diagnosis
* Verified sleep bruxism
* More than 18 Years
* Signed ICF

Exclusion Criteria:

* Contraindication of concomitant medication and diseases judged by investigator
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Reduction of number of grinds per hour per night | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Wendelboe, MsSc (Odont), Study Chair — Medotech A/S
Locations (1):
- Odontologisk Institute, Aarhus, Denmark